CLINICAL TRIAL: NCT01224132
Title: Effect of Probiotics in the Treatment of Children With Atopic Dermatitis
Brief Title: Effect of Probiotics in the Atopic Dermatitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Yuzuncu Yıl of the University Rector's Office of Scientific Research Department, Yuzuncu Yıl of the University Rector's Office of Scientific Research Department
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: JID-2010-0484
Record Dates: First submitted 2010-10-18; First posted 2010-10-19 (Estimated); Last update posted 2010-10-19 (Estimated); Status verified 2008-05

CONDITIONS: Atopic Dermatitis, Probiotics
Keywords: Atopic dermatitis, probiotic, SCORAD index, prick tests, cytokines
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotics (No Intervention)
  Interventions: Drug: probiotic ® pur
- skim milk powder, dextrose (No Intervention)
  Interventions: Drug: probiotic ® pur

INTERVENTIONS:
Drug: probiotic ® pur — daily, four types of probiotic bacteria ( Bifidobacterium bifidity, Lactobacillus acidophilus, Lactobacillus casei and Lactobacillus salivarium) 2 bags (two billion bacteria) (probiotic ® pur) for a total of 8 (eight) weeks

SUMMARY:
This study was designed to evaluate the efficacy of probiotics in the treatment of atopic dermatitis. Probiotics in AD patients were effective in reducing SCORAD index levels, but not effective in skin prick test positivity, serum IL-2-4-5-6-10, TNF-α, IFN-γ, ECP, and serum total and specific IgE levels.

DETAILED DESCRIPTION:
Frequently encountered in clinical practice, in the last 30 years, the prevalence of AD has rapidly increased as a result of industrialization. Thus, a new wave of quests for the treatment and prevention of AD has pushed forward. For the randomized, double-blinded, and placebo-controlled study this study was designed to evaluate the efficacy of probiotics in the treatment of AD. SCORAD positivity index of decline rates decline rates of the probiotic group of patients after treatment and skin prick tests were higher than that of the control group. While serum levels of IL-2-4-5-6-10, TNF-α, IFN-γ, ECP decreased in the probiotic group, only levels of IL-2-4-5, TNF-α decreased in the control group. The IgE decrease rate, the skin prick test, the serum total and specific of the probiotic group showed no difference from those of the control group. Probiotics in AD patients were effective in reducing SCORAD index levels, but not effective in skin prick test positivity, serum IL-2-4-5-6-10, TNF-α, IFN-γ, ECP, and serum total and specific IgE levels.

ELIGIBILITY:
Inclusion Criteria:SCORAD (SCORing Atopic Dermatitis) index is based on medium-heavy (Carr 2006). Age range is 1-13 with no patient showing evidence of any other disease except the existent disease -

Exclusion Criteria:No drug was used for 14 (fourteen) days prior to study, including antihistamines and steroids. Also, no occurrence of malabsorption, such as gastrointestinal disease, was detected.

-

Ages: 8 Weeks to 8 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2007-10; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)